CLINICAL TRIAL: NCT03720093
Title: Exploratory Analysis of Pulmonary Microbiome in Patients Intubated for Non-pulmonary Conditions- A Pilot Study
Brief Title: Exploratory Analysis of Pulmonary Microbiome in Intubated Patients
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Niguarda Hospital (Other); Parma University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Microbiota Polmonare in ICU
Record Dates: First submitted 2018-10-09; First posted 2018-10-25 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Intubation Complication
Keywords: ventilation; intubation; pulmonary microbiome
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, multicentric study investigates the modifications of pulmonary microbiome that occur in patients who need mechanical ventilation for non-pulmonary conditions. Genomic analysis will be performed by 16S RNA amplification on biological samples (bronchial aspirate) collected from patients.

DETAILED DESCRIPTION:
The microbiome is defined as a community of microorganisms (such as bacteria, fungi, and viruses) that inhabit a particular organ. This prospective, multicentric, observational study investigates the bacterial changes that occur in the pulmonary microbiome during the first 72 hours of mechanical ventilation in patients who have been intubated for non-pulmonary conditions in intensive care units (ICU).

To this aim, genetic analyses will be performed on bronchial aspirate samples that will be collected from patients during their staying in ICU. Demographic and clinical information will be retrieved from patients' clinical reports and recorded in an apposite clinical report forms (CRF) in anonymized way. In particular, the reason for the admission to ICU, absence fo concomitant pulmonary diseases, comorbidities, body mass index, hematological examination results, concomitant therapies, antibiotic therapy performed in the 30 days prior to the admission, ventilation associated pneumonia (VAP)-preventing procedures, complications during mechanical ventilation, length of mechanical ventilation will be recorded in the CRF.

The study will last 24 months.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo mechanical ventilation for non-pulmonary conditions (i.e. neurological condition)
* patients who are expected to need mechanical ventilation for >48 hours

Exclusion Criteria:

* diagnosis at the ICU admission of pneumonia
* need of mechanical ventilation for pulmonary conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients with mechanical ventilation for at least 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Changes of pulmonary microbiome between the time of intubation and 72 hours post-intubation, through genetic analysis of bacterial 16 Svedberg (16S) ribosomal RNA in bronchial aspirate. | At the time of intubation and after 72 hours from intubation
  Two samples of bronchial aspirate were collected (one at the time of incubation and one 72 hours post-intubation) and analyzed by Polymerase Chain Reaction (PCR) by amplifying 16 Svedberg (16S) ribosomal RNA. Primers that specifically recognize hypervariable regions of 16S sub-unit will be used. At 5' end an adaptor will be inserted to prepare the MiSeqsequencing library. The classification of microbiome taxa will be expressed as diversity measure (diversity index alpha or beta); the frequency of the most represented taxa and the confidence interval will be calculated. Differences in microbiome composition will be represented with the analysis of principal coordinates (PCoA) based on phylogenetic distance (matrix UNIFRAC).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, Professor, Study Director — University of Milano Bicocca; Andrea Gori, Professor, Study Chair — Fondazione Cà Granda, Policlinico Milano
Locations (3):
- Italy (3):
  - ASST-Monza, Monza, MB
  - Ospedale Niguarda, Milan
  - Ospedale di Parma, Parma

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be shared upon written request to the study director

REFERENCES:
- [Background] McDonald D, Ackermann G, Khailova L, Baird C, Heyland D, Kozar R, Lemieux M, Derenski K, King J, Vis-Kampen C, Knight R, Wischmeyer PE. Extreme Dysbiosis of the Microbiome in Critical Illness. mSphere. 2016 Aug 31;1(4):e00199-16. doi: 10.1128/mSphere.00199-16. eCollection 2016 Jul-Aug. PMID 27602409
- [Background] Zaborin A, Smith D, Garfield K, Quensen J, Shakhsheer B, Kade M, Tirrell M, Tiedje J, Gilbert JA, Zaborina O, Alverdy JC. Membership and behavior of ultra-low-diversity pathogen communities present in the gut of humans during prolonged critical illness. mBio. 2014 Sep 23;5(5):e01361-14. doi: 10.1128/mBio.01361-14. PMID 25249279
- [Background] Ojima M, Motooka D, Shimizu K, Gotoh K, Shintani A, Yoshiya K, Nakamura S, Ogura H, Iida T, Shimazu T. Metagenomic Analysis Reveals Dynamic Changes of Whole Gut Microbiota in the Acute Phase of Intensive Care Unit Patients. Dig Dis Sci. 2016 Jun;61(6):1628-34. doi: 10.1007/s10620-015-4011-3. Epub 2015 Dec 29. PMID 26715502
- [Background] Charlson ES, Bittinger K, Haas AR, Fitzgerald AS, Frank I, Yadav A, Bushman FD, Collman RG. Topographical continuity of bacterial populations in the healthy human respiratory tract. Am J Respir Crit Care Med. 2011 Oct 15;184(8):957-63. doi: 10.1164/rccm.201104-0655OC. Epub 2011 Jun 16. PMID 21680950
- [Background] Morris A, Beck JM, Schloss PD, Campbell TB, Crothers K, Curtis JL, Flores SC, Fontenot AP, Ghedin E, Huang L, Jablonski K, Kleerup E, Lynch SV, Sodergren E, Twigg H, Young VB, Bassis CM, Venkataraman A, Schmidt TM, Weinstock GM; Lung HIV Microbiome Project. Comparison of the respiratory microbiome in healthy nonsmokers and smokers. Am J Respir Crit Care Med. 2013 May 15;187(10):1067-75. doi: 10.1164/rccm.201210-1913OC. PMID 23491408
- [Background] Segal LN, Alekseyenko AV, Clemente JC, Kulkarni R, Wu B, Gao Z, Chen H, Berger KI, Goldring RM, Rom WN, Blaser MJ, Weiden MD. Enrichment of lung microbiome with supraglottic taxa is associated with increased pulmonary inflammation. Microbiome. 2013 Jul 1;1(1):19. doi: 10.1186/2049-2618-1-19. PMID 24450871
- [Background] Segal LN, Rom WN, Weiden MD. Lung microbiome for clinicians. New discoveries about bugs in healthy and diseased lungs. Ann Am Thorac Soc. 2014 Jan;11(1):108-16. doi: 10.1513/AnnalsATS.201310-339FR. PMID 24460444
- [Background] Berdal JE, Bjornholt J, Blomfeldt A, Smith-Erichsen N, Bukholm G. Patterns and dynamics of airway colonisation in mechanically-ventilated patients. Clin Microbiol Infect. 2007 May;13(5):476-80. doi: 10.1111/j.1469-0691.2006.01678.x. PMID 17430338